CLINICAL TRIAL: NCT04125030
Title: Instruments Validation and Correlational Explorations Between Clinical Recovery and Personal Recovery for the Evaluation of a Brief Intervention by Peer Support Workers in the Province of Quebec, Canada
Brief Title: Convergent and Concurrent Validity Between Clinical Recovery and Personal-civic Recovery in Mental Health
Status: Suspended | Type: Observational
Why Stopped: COVID-19 pandemic
Sponsor: Centre de Recherche de l'Institut Universitaire en santé Mentale de Montréal (Other)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Jean-Francois Pelletier, Principal Investigator, Centre de Recherche de l'Institut Universitaire en santé Mentale de Montréal
Other Study IDs: 2020-1948
Record Dates: First submitted 2019-10-08; First posted 2019-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Psychotic Disorders; Mood Disorders
MeSH Terms: conditions — Psychotic Disorders; Mood Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Validation of questionnaires — Participants will complete i) the RAS (24 items, 5-point Likert scale), ii) the CM (23 items, 5-point Likert scale), and the iii) the RSA for consumers (32 items, 5-point Likert scale). These participants have already completed these other measures (clinical recovery): iv-Anxiety: Anxiety State-Trait Anxiety Inventory Form Y6 (STAI-Y6) (6 items); v- Depression: Depression Patient Health Questionnaire (PHQ-9) (9 items) ; vi- Alcohol Dependence: Alcohol Use Disorders Identification Test (AUDIT-10) (10 items) ; vii- Drug Dependence: Drug Abuse Screening Test (DAST-10) (10 items) ; viii- Psychosis : Psychosis Screening Questionnaire (PSQ 12 items) ; ix- Social functioning : World Health Organization Disability Assessment Schedule (WHODAS 2.0) (12 items).

SUMMARY:
Several instruments have been developed by clinicians and academics specialized in mental health and psychiatry to assess clinical recovery in terms of symptom reduction. Based on their life narratives, measurement tools have also been developed and validated through participatory research programs by persons living with mental health problems or illnesses to assess a more personal experience of recovery as a way of leaving a meaningful and satisfying life despite and beyond ongoing disorders and symptoms of mental illness. Other instruments have also been developed to assess the degree to which mental health and psychiatric institutions are recovery-oriented. The overall aim of this project is to explore correlations between clinical recovery, personal recovery and this latter organizational recovery.

DETAILED DESCRIPTION:
The "signatures" of mental health problems or illnesses (MHPIs) is a term formulated by the National Institute of Mental Health (NIMH) to designate the broad range of genetic, biological, psychological, and social factors that may "sign" a specific mental disorder, depending on an individual's sex, history, lifestyle habits, and so on. In 2010, the Research Center of the Mental Health University Institute of Montreal (IUSMM) decided to develop the "Signature Bank" project for the collection of biological and dimensional signatures from all patients with MHPIs of the IUSMM (catchment area of about 600,000 inhabitants). Over 4,000 patients are treated annually at the IUSMM, while an additional 2,000 patients per year are treated by means of outpatient or ambulatory services. These activities provide us with one of the largest populations of psychiatric patients in Canada. This research project is based on the extensive involvement of the IUSMM-hospital site in the attempt to establish an exclusive niche for discoveries in the signatures of mental illnesses. By collaborating with the Research Centre, IUSMM-hospital managers have contributed to the implementation of this large-scale project that aims at measuring the genetic, biological, psychological, and social signatures of people living with MHPIs who use the IUSMM-hospital's clinical services, and who consent to taking part in this longitudinal research initiative. The goal of is study is to better understand not only the signatures of MHPIs, but that of recovery in mental health, and as reported by patients living with psychiatric disorders who will additionally fill out the French Recovery Assessment Scale (RAS), Recovery Self-Assessment (RSA) and Citizenship Measure (CM). Participants in the Signature Bank are routinely approached and recruited by a Research Nurse at their admission to the Psychiatric Emergency Department (T1) of the IUSMM. As of March 2019, 1862 eligible participants from the psychiatric emergency of the IUSMM have been approached. Of this number, 1218 agreed to participate and thus completed at least T1 of the Signature study. For all participants, the same measures are repeated at discharge (T2), at the first follow up at an outpatient clinic (T3), and finally (T4) when treatment ends or 12 months after T3. Our sample is characterized by individuals with psychotic disorders (N=166), or mood disorders (N=186), for a total of 352 patients who completed T3 and/or T4. All participants signed a detailed consent form, and the study was approved by the local ethics committee in accordance with the Declaration of Helsinki. Research Nurses collected patient's psychiatric diagnoses from medical records. They were established by psychiatrists on the ward, and coded according to the World Health Organisation International Classification of Disease (ICD-10). This study will use 2 of the categories of mental or behavioural disorder (F00-F99): 1) Schizophrenia and psychotic disorders (F20-F29), and 2) Mood disorders (F30-F39) who have enrolled in the Signature Bank for longitudinal studies and who have thus already completed questionnaires for clinical evaluation purposes (clinical recovery). Those who accept to participate in this study will further complete the RAS, the CM, and the RSA, which was developed to gauge the degree to which programs implement recovery-oriented practices and to identify strengths and areas of improvement as agencies strive to offer recovery-oriented care. Two specific research objectives are pursued. Firstly: measuring correlational relations between dimensions of personal recovery (RAS and CM), and levels of anxiety, depression, dependence, psychosis, and social functioning (clinical recovery). Secondly: validation of the psychometric properties of the French version of the RSA (organizational recovery). Statistical analyses will be performed to determine internal consistency (Cronbach alphas for each of the subscales), and construct validity (confirmatory or exploratory factor analyzes). Our power calculation has determined that 200 participants will be needed to test measurement invariance for sex and main psychiatric diagnosis (psychotic or mood disorders) in order to detect significant correlations with a Type I error of 5% and a power of 80%. Signature Bank participants will be contacted to complete i) the RAS (24 items, 5-point Likert scale), ii) the CM (23 items, 5-point Likert scale), and the iii) the RSA for consumers (32 items, 5-point Likert scale). These participants have already completed these other measures (clinical recovery): iv-Anxiety: Anxiety State-Trait Anxiety Inventory Form Y6 (STAI-Y6) (6 items); v- Depression: Depression Patient Health Questionnaire (PHQ-9) (9 items) ; vi- Alcohol Dependence: Alcohol Use Disorders Identification Test (AUDIT-10) (10 items) ; vii- Drug Dependence: Drug Abuse Screening Test (DAST-10) (10 items) ; viii- Psychosis : Psychosis Screening Questionnaire (PSQ 12 items) ; ix- Social functioning : World Health Organization Disability Assessment Schedule (WHODAS 2.0) (12 items).

Each patient diagnosed with F20-F39 disorders and who have completed at least T2 will be contacted by phone and asked to additionally fill out the RSA, RAS and CM. Those who will accept to be contacted will be invited to come to the IUSMM where they will be met by a Research Assistant. They will first read and sign the additional Information and Consent Form specific to this study or ask further questions before doing so. Secondly, they will fill out the RSA, RAS and CM on a touch screen device. Data will be stored on the Signature Bank secured server. If necessary, future new participants who will have completed T2 will be contacted in the same way until the required number of participants is reached. There are typically 60 to 80 new participants per month to the Signature Bank. Test-retest reliability will be investigated, as well as internal consistency, construct validity of these RSA, RAS and CM tools, correlations between their subscales and those of anxiety, depression, substance misuse, psychosis, and social functioning measures, in and across psychiatric diagnoses, and sex. The same i-iv measures will be used in a future project to assess the effect of a brief intervention by Peer Support Workers (PSW) with a control group. A Randomized Control Trial with future IUSMM patients who will have accepted to be enrolled in the Signature Bank will be proposed to compare treatment as usual to treatment as usual plus the PSW intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participants of the Signature Bank who completed at least T2.

Exclusion Criteria:

* Patients with learning disabilities

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Patients diagnosed with schizophrenia and psychotic disorders
  * Patients diagnosed with Mood disorders
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of patients' current status : anxiety (clinical recovery) | 9 months
  Participating patients will fill out the Anxiety State-Trait Anxiety Inventory Form Y6 (STAI-Y6). This is a 6-item questionnaire with 4-point Likert scales (1-2-3-4). Higher scores are positively correlated with higher levels of anxiety. Minimum score = 6 : maximum score = 24.
  Data will be aggregated for statistical analyses (convergent validation and confirmatory factor analyses) and measurement of invariance for sex (male/female) and main psychiatric diagnosis (psychotic/mood disorders).
Assessment of patients' current status : depression (clinical recovery) | 9 months
  Participating patients will fill out the Depression Patient Health Questionnaire (PHQ-9). This is a 9-item questionnaire with 4-point Likert scales (0-1-2-3). Higher scores are positively correlated with higher levels of depression. Minimum score = 0 : maximum score = 27.
  Data will be aggregated for statistical analyses (convergent validation and confirmatory factor analyses) and measurement of invariance for sex (male/female) and main psychiatric diagnosis (psychotic/mood disorders).
Assessment of patients' current status : alcohol dependence (clinical recovery) | 9 months
  Participating patients will fill out the Alcohol Use Disorders Identification Test (AUDIT-10). This is a 10-item questionnaire with 5-point Likert scales (0-1-2-3-4). Higher scores are positively correlated with higher levels of alcohol dependence. Minimum score = 0 : maximum score = 40.
  Data will be aggregated for statistical analyses (convergent validation and confirmatory factor analyses) and measurement of invariance for sex (male/female) and main psychiatric diagnosis (psychotic/mood disorders).
Assessment of patients' current status : drug dependence (clinical recovery) | 9 months
  Participating patients will fill out the Drug Abuse Screening Test (DAST-10). This is a 10-item questionnaire with no-yes answers (0-1). Higher scores are positively correlated with higher levels of drog dependence. Minimum score = 0 : maximum score = 10.
  Data will be aggregated for statistical analyses (convergent validation and confirmatory factor analyses) and measurement of invariance for sex (male/female) and main psychiatric diagnosis (psychotic/mood disorders).
Assessment of patients' current status : psychosis (clinical recovery) | 9 months
  Psychosis Screening Questionnaire (PSQ 12 items) with no-unsure-yes answers (1-2-3). Higher scores are positively correlated with higher levels of psychosis. Minimum score = 12 : maximum score = 36.
  Data will be aggregated for statistical analyses (convergent validation and confirmatory factor analyses) and measurement of invariance for sex (male/female) and main psychiatric diagnosis (psychotic/mood disorders).
Assessment of patients' current status : social functioning (clinical recovery) | 9 months
  Participating patients will fill out the World Health Organization Disability Assessment Schedule (WHODAS 2.0). This is a 12-item questionnaire with 5-point Likert scales (0-1-2-3-4). Lower scores are positively correlated with higher levels of social functioning. Minimum score = 0 : maximum score = 48.
  Data will be aggregated for statistical analyses (convergent validation and confirmatory factor analyses) and measurement of invariance for sex (male/female) and main psychiatric diagnosis (psychotic/mood disorders).
Assessment of patients' current status : recovery (personal recovery) | 9 months
  Participating patients will fill out the Recovery Assesment Scale (RAS). This is a 24-item questionnaire with 5-point Likert scales (1-2-3-4-5). Higher scores are positively correlated with higher levels of recovery. Minimum score = 24 : maximum score = 120.
  Data will be aggregated for statistical analyses (convergent validation and confirmatory factor analyses) and measurement of invariance for sex (male/female) and main psychiatric diagnosis (psychotic/mood disorders).
Assessment of patients' current status : citizenship (personal recovery) | 9 months
  Participating patients will fill out the Citizenship Measure (CM). This is a 23-item questionnaire with 5-point Likert scales (1-2-3-4-5). Higher scores are positively correlated with higher levels of citizenship. Minimum score = 23 : maximum score = 115.
  Data will be aggregated for statistical analyses (convergent validation and confirmatory factor analyses) and measurement of invariance for sex (male/female) and main psychiatric diagnosis (psychotic/mood disorders).

SECONDARY OUTCOMES:
Patient Experience : organizational recovery | 9 months
  Participating patients will fill out the Recovery Self-Assessment (RSA-for consumers), to assess their current experience of mental healthcare. This tool was developed to gauge the degree to which programs implement recovery-oriented practices and to identify strengths and areas of improvement as agencies strive to offer recovery-oriented care. This is a 32-item questionnaire with 5-point Likert scales (1-2-3-4-5). Higher scores are positively correlated with higher levels of recovery-oriented care. Minimum score = 32 : maximum score = 160.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Pelletier, PhD, Principal Investigator — IUSMM Research Centre
Locations (1):
- CR-IUSMM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pelletier JF, Corbiere M, Lecomte T, Briand C, Corrigan P, Davidson L, Rowe M. Citizenship and recovery: two intertwined concepts for civic-recovery. BMC Psychiatry. 2015 Mar 4;15:37. doi: 10.1186/s12888-015-0420-2. PMID 25885779